CLINICAL TRIAL: NCT05077813
Title: Utilizing the Crosstalk Among Chicoric Acid, 13-Cis Retinoic Acid(Aerosolized), Minocycline and Vitamin D as a Potent Quadrate Therapy for Treating Patients With Multidrug-resistant TB and Patient With Both Multidrug-resistant TB and COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Collaborators: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Mahmoud Ramadan mohamed Elkazzaz, Clinical Scientist, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: How to kill Tuberculosis
Record Dates: First submitted 2021-10-10; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Isotretinoin; Minocycline; Vitamin D; Alitretinoin; Tretinoin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 13 cis retinoic acid, Minocycline, Chicroic Acid and Vitamin D for (MDR-TB) (Active Comparator): 50 Subjects will be randomly assigned to receive A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized 13 cis retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets contain choric acid = 3.4 to 8.5 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Interventions: Combination Product: 13 cis retinoic acid, Minocycline, Chicroic Acid and Vitamin D for (MDR-TB)
- 9 cis retinoic acid , Minocycline,Chicroic Acid and Vitamin D for (MDR-TB) (Active Comparator): 50 Subjects will be randomly assigned to receive A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized 9 cis retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets contain choric acid = 3.4 to 8.5 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Interventions: Combination Product: 9 cis retinoic acid, Minocycline, Chicroic Acid and Vitamin D for (MDR-TB)
- All trans retinoic acid , Minocycline,Chicroic Acid and Vitamin D for (MDR-TB) (Active Comparator): 50 Subjects will be randomly assigned to receive A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized All trans retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets contain choric acid = 3.4 to 8.5 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Interventions: Combination Product: All trans retinoic acid , Minocycline,Chicroic Acid and Vitamin D for (MDR-TB)
- 13 cis retinoic acid, Minocycline, Chicroic Acid and Vitamin D For (COVID-19 and MDR-TB) (Active Comparator): 50 Subjects with confection of COVID-19 and multidrug-resistant tuberculosis (MDR-TB) will be randomly assigned to receive A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized 13 cis retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets contain choric acid = 3.4 to 8.5 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Interventions: Combination Product: 13 cis retinoic acid, Minocycline, Chicroic Acid and Vitamin D For (COVID-19 and MDR-TB)
- All trans retinoic acid, Minocycline, Chicroic Acid and Vitamin D For (COVID-19 and MDR-TB) (Active Comparator): 50 Subjects with confection of COVID-19 and multidrug-resistant tuberculosis (MDR-TB) will be randomly assigned to receive A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized All trans retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets contain choric acid = 3.4 to 8.5 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Interventions: Combination Product: All trans retinoic acid, Minocycline, Chicroic Acid and Vitamin D For (COVID-19 and MDR-TB)
- The standard therapy (Placebo Comparator): The standard therapy 100 infected patients with confection of COVID-19 and MDR-TB will receive the standard therapy for tuberculosis for 30 days 50- 50-
  Interventions: Other: The standard therapy

INTERVENTIONS:
Combination Product: 13 cis retinoic acid, Minocycline, Chicroic Acid and Vitamin D for (MDR-TB) — A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized 13 cis retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets contain choric acid = 3.4 to 8.5 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Arms: 13 cis retinoic acid, Minocycline, Chicroic Acid and Vitamin D for (MDR-TB)
Combination Product: 9 cis retinoic acid, Minocycline, Chicroic Acid and Vitamin D for (MDR-TB) — A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized 9 cis retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets contain choric acid = 3.4 to 8.5 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Arms: 9 cis retinoic acid , Minocycline,Chicroic Acid and Vitamin D for (MDR-TB)
Combination Product: All trans retinoic acid , Minocycline,Chicroic Acid and Vitamin D for (MDR-TB) — Active Comparator: All trans retinoic acid , Minocycline,Chicroic Acid and Vitamin D 50 Subjects will be randomly assigned to receive A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized All trans retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets contain choric acid = 3.4 to 8.5 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Arms: All trans retinoic acid , Minocycline,Chicroic Acid and Vitamin D for (MDR-TB)
Combination Product: All trans retinoic acid, Minocycline, Chicroic Acid and Vitamin D For (COVID-19 and MDR-TB) — 50 Subjects with confection of COVID-19 and multidrug-resistant tuberculosis (MDR-TB) will be randomly assigned to receive A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized All trans retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets contain choric acid = 3.4 to 8.5 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Arms: All trans retinoic acid, Minocycline, Chicroic Acid and Vitamin D For (COVID-19 and MDR-TB)
Combination Product: 13 cis retinoic acid, Minocycline, Chicroic Acid and Vitamin D For (COVID-19 and MDR-TB) — 50 Subjects with confection of COVID-19 and multidrug-resistant tuberculosis (MDR-TB) will be randomly assigned to receive A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized 13 cis retinoic acid in gradual 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets contain choric acid = 3.4 to 8.5 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4
  Arms: 13 cis retinoic acid, Minocycline, Chicroic Acid and Vitamin D For (COVID-19 and MDR-TB)
Other: The standard therapy — The standard therapy 100 infected patients with confection of COVID-19 and MDR-TB will receive the standard therapy for tuberculosis for 30 days
  Arms: The standard therapy

SUMMARY:
Utilizing the Crosstalk Among Chicoric Acid, 13-Cis Retinoic Acid(Aerosolized), Minocycline and Vitamin D as a Potent Quadrate Therapy for treating patients with Multidrug-resistant TB and patient with both Multidrug-resistant TB and COVID-19 . A double-edged sword Clinical Study

I)Part of Tuberculosis

Tuberculosis (TB) is a major infectious disease killer globally. It affected 10 million and killed 1.4 million people in 2019 alone. The predicted impact of the COVID-19 pandemic is an additional 190,000 TB deaths in 2020, and it is expected in the next 5 y that there will be up to a 20% increase in the global TB disease burden , stressing the critical need for new safe and effective drugs against Mycobacterium tuberculosis (Mtb). In addition, controlling multidrug-resistant TB (MDR-TB) presents a huge public health challenge . New drug discovery could require several years with no guarantee but repurposing established may be useful to treat patients with tuberculosis . Here we demonstrate that we could utilize the crosstalk among Chicoric Acid, 13-Cis Retinoic Acid, Minocycline , and vitamin D as a novel quadrate therapy against TB.Drug-resistant tuberculosis represents a global emergency, requiring new drugs. Recently Minocycline was found to be highly potent in laboratory strains of Mycobacterium TB, and 30 drug-sensitive and multidrug/extensively drug-resistant clinical strains were susceptible to clinically attainable dosages. The lung concentration-time profiles of a 7 mg/kg/day human-equivalent minocycline dosage yielded bacterial kill rates comparable to first-line antituberculosis drugs. Extracellular bacilli were destroyed directly by minocycline. Minocycline also killed intracellular bacilli indirectly through granzyme A-driven apoptosis. Furthermore, minocycline showed dose-dependent antiinflammatory effect, suggesting that it may protect tuberculosis patients against immunopathology. A study showed that M. tuberculosis induced the expression of indoleamine 2,3-dioxygenase (IDO), an enzyme involved in tryptophan catabolism, in macrophages and in the lungs of animals (mice and macaque) with active disease. In a macaque model of inhalation TB, suppression of IDO activity reduced bacterial burden, pathology, and clinical signs of TB disease, leading to increased host survival. This increased protection was accompanied by increased lung T cell proliferation, induction of inducible bronchus-associated lymphoid tissue and correlates of bacterial killing . A recent study showed that Minocycline-induced significantly inhibition of IDO expression. But Minocycline-induced inhibition of IDO expression is retinoid-dependent. The combined treatment with minocycline and retinol, however, resulted in a striking, statistically significant decrease in IDO. Co-treatment with minocycline and retinol again resulted in decreased TNF-α and IL-6 levels. A study showed that IL-6 inhibits IFN-γ induced autophagy in Mycobacterium (TB) H37Rv infected macrophages. As well as neutralization of endogenous IL-6 by anti-IL-6 antibody significantly enhances the IFN-γ mediated killing of the intracellular bacteria. Minocycline's anti-inflammatory effects are mediated through RAR signaling. Therefore, The combined treatment with minocycline and retinol is expected to effectively inhibit (TB) and its inflammatory complication, Fortunately, Retinoic Acid significantly inhibits the in vivo growth of M. tuberculosis and the development of tuberculosis. In addition to, 13-Cis RA and Chicoric Acid ( CA ) enhanced the cell surface expression of HLA-DR and CD14 molecules on U937 macrophages and prevented the growth of Mtb within macrophages. Moreover, 13-cis RA and CA, have increased NO generation compared to untreated control macrophages, significantly . Both drugs have a significant inhibitory effect on Mtb growth but CA at the highest concentration was more potent than 13-cis RA . Therefore we will use retinoic acid to induce the effect of Minocycline as well as its ability to inhibit tuberculosis in combination with CA .Recent data showed that Vitamin D support innate immune responses to Mycobacterium TB and Low vitamin D levels were associated with a 5-fold increased risk for progression to tuberculosis. Deficiency of vitamin D has long been implicated in activation of (TB) . Serum vitamin D in TB patients are lower than in healthy controls . Vitamin D has been found to speed up the clearance of (TB) bacteria from the lungs of people with multi-drug resistant TB, according to a study of 1,850 patients. It was showed that Vitamin D receptor (VDR) must form a heterodimer complex with retinoid X receptor (RXR) to regulate gene transcription. Retinol plays a crucial role in lung development and signaling the vitamin D pathway. 9-cis-retinoic acid, an active vitamin A metabolite and the ligand of RXR, assists VDR signaling and suppresses the degradation of circulating vitamin D.

DETAILED DESCRIPTION:
This double blinded, randomized, placebo controlled trial on the clinical efficacy and antimicrobial mechanisms of quadrate therapy(Chicoric Acid, 13-Cis Retinoic Acid(Aerosolized), Minocycline and Vitamin D) as a Potent Quadrate Therapy Against Tuberculosis. 200 men and women will be enrolled , who are age 18 to 65 years inclusive, have at least two positive sputum smears for tuberculosis (TB), and have given informed consent to participate in the study. All of the enrollees will have active TB . The effect of the quadrate therapy status will be examined in the context of a randomized trial conducted in Egyptian or Saudi Arabian Subjects will be randomized to receive either the quadrate therapy or placebo from the start of their TB therapy, through the 1 months of anti-TB therapy, and until the last recruited patient reaches 6 months of follow up. Thus, the first subject is likely to be followed for 12 months, assuming the duration of recruitment is 12 months. The endpoints of interest include bacteriologic cure, immune response parameters, and clinical outcomes. The researchers will also examine the utility of these immune response parameters as surrogate markers for treatment efficacy in TB, irrespective of the quadrate therapy and other risk factors. The study will be carried out as a collaborative effort between. Kafr elshiekh university ,Faculty of Medicine, Egypt and First health cluster ,Ministry of health ,Saudia Arabia. Subjects will be randomly assigned to receive A) Minocycline i.v. 4,5 mg/kg gradual in 2 divided doses increases from 4,5 mg/kg from the first week to 7.5 and 10 mg/kg to the last week. In addition to Aerosolized 13 cis retinoic acid or All trans retinoic acid or 9 cis retinoic acid gradual in 2 divided doses increases from 0.2 mg/kg/day to 4 mg/kg/day as inhaled retinoic acid therapy for 30 days. Moreover, the patients will receive Echinacea Purpurea Extract Capsules Polyphenols Chicoric Acid .Chicoric acid (also known as cichoric acid and dicaffeoyltar- taric acid) is the main phenolic compound found in Echinacea purpurea. Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. Each batch of tablets Caffeic acid derivative levels are typically as follows: caftaric acid = 0.5 to 2.0 mg/tablet; cichoric acid = 3.4 to 8.5 mg/tablet; chlorogenic acid = < 0.5 mg/tablet; dicaffeoyl quinic acids (including cynarin) = 0.7 to 2.0 mg/tablet; echinacoside = 1.0 to 1.7 mg/tablet. Furthermore, the patients will receive Cholecalciferol(Vitamin D) Intramuscular injection of 600,000 units of Cholecalciferol for 2 doses given at week 0 and week 4 (b) placebo. The primary objectives are to: (1) determine the efficacy of the quadrate therapy on sputum and culture negativity at one month and two months; (2) determine the efficacy of micronutrient supplements on survival between two arms at 8 and 24 months; and (3) determine the efficacy of micronutrient supplements on TB relapse and reinfection. Secondary study objectives are to: (1) compare the treatment arms with respect to absolute change in CD4 counts from 0 to 1, 6, 12 months; (2) compare the treatment arms with respect to weight change from baseline and1 months, 6 months, and 12 months; (3) compare the treatment arms with respect to immunological parameters, namely ex vivo lymphocyte proliferation; and cytokine production, namely IL-2, IL-6, INF-g INF-Alpha, IL-12, and TNF-a, and Interferon alpha at 1, 6, 12 months; and (4) correlate the above mentioned immunological markers with smear conversion rates at 1 month, 2 months, cure, relapse, and death. Finally, we suggest that this combination therapy will effectively inhibit tuberculosis infection and achieve treatment with significant effect against (TB)

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 up to 65 years
* Microbiologically or histologically confirmed active tuberculosis as well as confirmed positive with COVID-19
* Clinically confirmed latent tuberculosis
* Drug resistant MTb
* Negative pregnancy test for 18-40 year-old females
* Able to sign consent

Exclusion Criteria:

* HIV positive
* Known intolerance of vitamin D
* Sarcoidosis
* Hyperparathyroidism or nephrolithiasis
* Taking vitamin D or A supplementation in the two months preceding enrolment
* Baseline serum corrected calcium >2.65 mmol/L
* Current haemodialysis
* Children, pregnant or breastfeeding individuals
* Concomitant benzothiadiazine derivative, cardiac glycoside, carbamazepine, phenobarbital, phenytoin, primidone or long-term immunosuppressant therap
* Extra-pulmonary or smear negative tuberculosis
* Patients receiving steroids, cytotoxic drugs, post transplant or metastatic malignancy, or not expected to survive for the duration of ATT
* Pregnant or lactating women
* Active diarrhoea, indicating possible fat-soluble vitamin malabsorption.
* Baseline Hypercalcemia >10.5 mg/dl
* Concurrent use of cyclosporin, cisplatin, amfotericin B, cephalosporins, polymyxins and vancomycin.
* History of adverse events on previous Minocycline or other tetracycline use (by spontaneous reporting nor by active questioning).
* Depressive disorder
* Body mass index less than 18 points or higher than 25 points
* Contraindications for hormonal contraception or intrauterine device.
* Autoimmune diseases A history of organ, bone marrow or hematopoietic stem cell transplantation
* Patients receiving anti-hcv treatment
* Permanent blindness in one eye
* History of iritis, endophthalmitis, scleral inflammation or retinitis 15-90 days of retinal detachment or eye surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Time to first negative SARS-CoV-2 PCR in NP swap and Mycobacterium tuberculosis sputum culture | within 4 weeks

SECONDARY OUTCOMES:
Sputum culture result (positive or negative)& COVID-19 PCR (positive or negative) | 2 weeks after therapy start date
Serum levels of CRP and ESR | one month
All cause mortality rate | one month
Absolute lymphocyte counts (CD4,CD8 and CD25+FOXP3+ Regulatory T) | one month
Measurement of cytokine (IFN-gamma and alpha , IL-6, IL-10, TNF-alpha, TGF-beta) levels produced in response to M. tb. | one month
Vitamin D status | one month
  Serum 25(OH)D concentrations
Retinoic acid status | one month
  Serum Retinoic acid concentrations
Minocycline status | one month
  Serum Minocycline concentrations
Serum indoleamine 2,3-dioxygenase (IDO) enzyme status | one month
  Serum indoleamine 2,3-dioxygenase (IDO) enzyme concentration
Chicoric Acid status | one month
  Serum Chicoric Acid concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mahmoud R Elkazzaz, M.Sc of Biochemistry, Principal Investigator — Faculty of Science , Damietta University; Amr K Ahmed, Principal Investigator — Ministry of Health
Locations (2):
- Kafr El-sheikh University, Cairo, Kafr el-Sheikh Governorate, Egypt
- Ministry of health. First health cluster, Riyadh, Riaydh, Saudi Arabia